CLINICAL TRIAL: NCT05585983
Title: INfluenza VaccInation To Mitigate typE 1 Diabetes (INVITED Trial)
Brief Title: INfluenza VaccInation To Mitigate typE 1 Diabetes
Acronym: INVITED
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ole Frøbert, MD, PhD, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INVITED-2022
Record Dates: First submitted 2022-10-15; First posted 2022-10-19 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: In this double blind, placebo-controlled clinical trial participants are allocated to either influanza vaccination (active) or to placebo (control).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The following are masked in the study: Participant, Care Provider, Investigator, Outcomes Assessor.
  The following are not masked: unblinded study nurses at participating sites randomizing participants in the eCRF system. The unblinded study nurses are not otherwise involved or participating in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Influenza vaccination (Experimental): Influenza vaccine, 0.5 mL.
  Interventions: Biological: Vaxigrip Tetra Sanofi Pasteur Europe
- Placebo (Placebo Comparator): Placebo, 0.5 mL saline.
  Interventions: Biological: Vaxigrip Tetra Sanofi Pasteur Europe

INTERVENTIONS:
Biological: Vaxigrip Tetra Sanofi Pasteur Europe — We will use 0.5 mL standard dose quadrivalent influenza vaccine containing 15 μg of hemagglutinin per strain consistent with WHO recommendations according to season.

SUMMARY:
In a multicenter, prospective, randomized, controlled clinical trial to compare influenza vaccination and placebo in sustaining β cell function in early type 1 diabetes mellitus.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is an autoimmune disease in which T cells attack and destroy the insulin-producing β cells in the pancreatic islets. In theory, immunotherapies aimed at re-programming the immune system to avoid β cell destruction is a promising strategy to prevent T1D or delay onset of overt disease.

In this trial we test the hypothesis that influenza vaccination is superior to no influenza vaccination in sustaining β cell function in early T1D. Secondary outcome measures include change in autoantibodies directed against antigens present in the pancreatic islets, measures of severity of disease, change in inflammatory markers, and antibody titers against the four viruses included in the vaccine.

Despite improvements in care, T1D is a leading cause of debilitating complications and early death globally. Children with residual β cell function are at lower risk for severe hypoglycemia, have better diabetes regulation, and have lower insulin requirements compared to children without residual β cell function. Thus, a simple, cheap treatment to mitigate T1D is highly warranted.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized with newly diagnosed type 1 diabetes mellitus.
* Written informed consent (parents, legal guardian).

Exclusion Criteria:

* Influenza vaccination during the current influenza season.
* Strong indication for influenza vaccination for non-diabetic disease.
* Severe allergy to eggs or previous allergic reaction to influenza vaccine.
* Suspicion of febrile illness or acute, ongoing infection.
* Hypersensitivity to the active substances or ingredients of Vaxigrip Tetra or against any residues, such as eggs (ovalbumin or chicken proteins), neomycin, formaldehyde and octoxinol.
* Patients with endogenic or iatrogenic immunosuppression that may result in reduced immunization response.
* Inability to provide informed consent from a parent or legal guardian.
* Age <7 or ≥18 years.
* Previous randomization in the INVITED trial.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in fasting residual β cell (C-peptide) function. | 12 months
  Measured as the area under the concentration-time curve (AUC) for mixed-meal tolerance test-stimulated C-peptide concentration over 4 hours relative to baseline (AUC 0-4 h, C-peptide, 12 months/ AUC 0-4 h, C-peptide, baseline)

SECONDARY OUTCOMES:
Change in fasting residual β cell (C-peptide) function. | 6 months.
  Measured as the area under the concentration-time curve (AUC) for mixed-meal tolerance test-stimulated C-peptide concentration over 4 hours relative to baseline (AUC 0-4 h, C-peptide, 6 months/ AUC 0-4 h, C-peptide, baseline)
Change in HbA1c | 12 months.
  Measured as standard laboratory test in mmol/mol
Change in insulin requirements. | 12 months.
  Measured as total insulin dose per kg body weight per day as a mean for the last 14 days.
Time-In-Range of blood glucose. | 12 months.
  Defined as percentage time in range (3.9-10.0 mmol/L) of continuous glucose monitoring over 14 days.
Variation of blood glucose. | 12 months.
  Determined as percent coefficient of variation of blood glucose over 14 days.

OTHER OUTCOMES:
Proportion of participants with stimulated C-peptide >0.2 pmol/mL | 12 months
  Proportion of participants in each of the treatment groups with stimulated C-peptide >0.2 pmol/mL
HbA1c time in range | 12 months.
  Defined as percentage time in range (48mmol/mol or below)
Insulin Dose Adjusted A1c | 12 months
  Defined as: IDAA1c = HbA1c (%) +4*total daily insulin dose (IE/kg/24 h)
Variation of blood glucose. | 6 months.
  Determined as percent coefficient of variation of blood glucose over 14 days.
Change in GAD 65 antibodies. | 12 months.
  Laboratory method to be determined
Change in GAD 65 antibodies. | 6 months.
  Laboratory method to be determined.
Change in regulatory T cells. | 12 months.
  Defined as percentage change.
Change in insulin autoantibodies. | 12 months.
  Laboratory method to be determined.
Change in zinc transporter-8 autoantibodies | 12 months.
  Laboratory method to be determined.
Change in islet cell autoantibodies. | 12 months.
  Laboratory method to be determined.
Change in cytokine levels. | 12 months.
  Markers to be determined: IL2, IL6, IL8, IL10, TNFα. Laboratory method to be determined.
Change in cytokine levels. | 6 months.
  Markers to be determined: IL2, IL6, IL8, IL10, TNFα. Laboratory method to be determined.
Unplanned hospitalizations. | 12 months.
  Number of unplanned hospitalizations with reasons for hospitalizations.
Serum hemagglutinin inhibition antibody titers against the four viruses included in the vaccine | 12 months.
  Antibody titers.
Serum hemagglutinin inhibition antibody titers against the four viruses included in the vaccine | 6 months.
  Antibody titers.
Clnical endpoints. | Up to 5 years.
  Hospitalizations and unplanned hospital contacts.
Treatment-emergent hypoglycemic events (safety outcome) | Up to 12 months.
  Hypoglycemic events reported according to the American Diabetes Association classification
Treatment-emergent events of diabetic ketoacidosis (safety outcome) | Up to 12 months.
  Events of diabetic ketoacidosis.

CONTACTS AND LOCATIONS:
Locations (10):
- Denmark (10):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Steno Diabetes Center Copenhagen, Copenhagen
  - Gødstrup Hospital, Herning
  - Holbaek Sygehus, Holbæk
  - Nykoebing F Sygehus, Nykøbing Falster
  - Randers Regional Hospital, Randers
  - Sjællands Universitetssygehus, Roskilde
  - Slagelse Hospital, Slagelse
  - Viborg Regional Hospital, Viborg

REFERENCES:
- [Derived] Pedersen IB, Kjolby M, Hjelholt AJ, Madsen M, Christensen AR, Adolfsen D, Hjelle JS, Kremke B, Stovring H, Jessen N, Vestergaard ET, Kristensen K, Frobert O. INfluenza VaccInation To mitigate typE 1 Diabetes (INVITED): a study protocol for a randomised, double-blind, placebo-controlled clinical trial in children and adolescents with recent-onset type 1 diabetes. BMJ Open. 2024 Jul 1;14(6):e084808. doi: 10.1136/bmjopen-2024-084808. PMID 38950997